CLINICAL TRIAL: NCT01785667
Title: Incidence of Retinopathy and Associated Risk Factors in Children and Young Adults With Type 1 Diabetes in Denmark
Acronym: DCPD1987
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Center for Eye Research Australia (Other); Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Rebecca Broe Pedersen, MD, Odense University Hospital
Other Study IDs: S-20100088
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Type 1 Diabetes; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Years
Biospecimen Retention: Samples With DNA — buffy coat, whole blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young Danish adults with type 1 diabetes: This is an observational study with no interventions.

SUMMARY:
The objective of this study is to clarify the current diabetic status, including development of complications, in a nationwide cohort of type 1 diabetics, who were last examined together in a large study in 1995. These youngsters were originally participating in a nationwide study of children with type 1 diabetes in Denmark back in 1986. The investigators will try to establish risk factors for developing diabetic retinopathy. The investigators will have emphasis on retinal vessel geometry and the possibilities for early detection of reversible retinal changes, and prediction of other vascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the follow-up study in 1995

Exclusion Criteria:

* No retinal photographs from 1995

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study includes a cohort of type 1 diabetic patients, who originally were identified in 21 paediatric departments and studied in 1986. This group initially consisted of 1033 children and was estimated to involve around 80 percent of all Danish type 1 diabetic patients below the age of 18. In 1995 further examinations were performed on the cohort; this time 339 chose to participate.
  In this study we will invite the participants from 1995 who also participated in the eye examinations, n=324, to participate in yet another follow-up examination.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Incidence of diabetic retinopathy and proliferative diabetic retinopathy | 16 years
  Using the ETDRS grading protocol the degree of retinopathy in 2011 will be assessed by grading 7-field fundus photographs taken at follow-up examination. This will be related to the degree of retinopathy found in the patients in 1995, where the last study of the cohort took place.

SECONDARY OUTCOMES:
Vessel diameters as a predictor of diabetic retinopathy and proliferative diabetic retinopathy | 16 years
  Using the computer software named IVAN we will assess the average vessel diameters around the optic disc on fundus photos from 1995. This we will relate to the degree of retinopathy in 2011 to see if vessel diameters predicts diabetic eye complications.

OTHER OUTCOMES:
Fractal dimensions as a predictor of diabetic retinopathy and proliferative diabetic retinopathy | 16 years
  Using the computer software named Fractal Analyzer we will assess the fractal dimension around the optic disc on fundus photos from 1995. This we will relate to the degree of retinopathy in 2011 to see if fractals can help predict diabetic eye complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Odense University Hospital, Odense, Fyn, Denmark